CLINICAL TRIAL: NCT01599169
Title: Evaluation of the Efficacy and Tolerance of B-Back® on the Burnout Syndrome. Double-blind, Randomized, Monocentric Trial With Two Parallel Groups (B-Back® Verum Versus B-Back® Placebo)
Brief Title: Evaluation of the Efficacy and Tolerance of B-Back® on the Burnout Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Collaborators: Nanox International Laboratory (Belgique) (Unknown)
Responsible Party: Principal Investigator, Alain Jacquet, MD, Université Victor Segalen Bordeaux 2
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ID-RCB : 2012 - A00096 - 37; e530 (Other: Clinical Pharmacology Department of University Victor Segalen Bordeaux 2)
Record Dates: First submitted 2012-05-06; First posted 2012-05-15 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Efficacy and Tolerance of B-Back® on the Burnout Syndrome
Keywords: Burnout syndrome; Depression work-related; Food supplement
MeSH Terms: conditions — Burnout, Psychological | interventions — Taurine; Siberian ginseng root; Extramel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B-Back® verum (Experimental)
  Interventions: Dietary Supplement: Dietary supplement : B-Back® (α-casozepine, taurine, eleutherococcus senticosus, Extramel)
- B-Back® placebo (Placebo Comparator)
  Interventions: Dietary Supplement: B-Back® placebo (without active compounds)

INTERVENTIONS:
Dietary Supplement: Dietary supplement : B-Back® (α-casozepine, taurine, eleutherococcus senticosus, Extramel) — 2 tablets/day after breakfast during 12 weeks
  Arms: B-Back® verum
Dietary Supplement: B-Back® placebo (without active compounds) — 2 tablets/day after breakfast during 12 weeks
  Arms: B-Back® placebo

SUMMARY:
The purpose of this study is to determine the efficacy and the tolerance of the food supplement B-Back®, containing α-casozepine, taurine, eleutherococcus senticosus and Extramel®, on the burnout syndrome.

DETAILED DESCRIPTION:
The burnout syndrome currently concern all the professional categories. In 2010 the WHO estimated that the three countries with the most important work-related depression are Unites States, Ukraine and France. The direct and indirect costs of work-related stress for the insurance program were not insignificant.

The purpose of this study is to determine the efficacy of the food supplement B-Back® proposed in order to improved the symptoms of the burnout syndrome : stress, fatigue, emotional imbalance, anxiety, sleep, etc.

The main objective is to determine the efficacy of B-Back® on the symptoms suggestive of the burnout syndrome by using the Burnout Measure Short version (BMS-10). The others objectives were to evaluate the tolerance of the product, to evaluate the efficacy of B-Back® on the symptoms suggestive of the burnout syndrome by using the Maslach Burnout Inventory, depression, and the global quality of professional and family life, sleep,and fatigue (energy).

ELIGIBILITY:
Inclusion Criteria:

* males and females outpatients aged 30-65 years old
* practicing professionals in contact with patients, students,...
* symptoms suggestive of burnout syndrome
* minimum score to the BMS-10 = 4
* able to understand the sdudy documents
* agreeing to go to dates of controls
* able to give informed consent
* affiliated to a French national insurance program

Exclusion Criteria:

* current anxiolytic or antidepressant treatment
* allergy known about one of the components of the food complement in the study
* intolerance in the lactose and in the proteins of milk
* pregnancy or feeding
* progressive pathology involving life-threatening during study
* professional on sick leave
* cancer not stabilized for at least five years or considered as not recovered
* subjects deprived of liberty court decision
* subjects in the psychic incapacity to understand the constraints of the study

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Burnout Measure Short version (BMS-10) score at 12 weeks | baseline and after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in BMS-10 score at 6 weeks | baseline and after 6 weeks
Change from baseline in Maslach Burnout Inventory score at 6 weeks | baseline and after 6 weeks
Change from baseline in Maslach Burnout Inventory score at 12 weeks | baseline and after 12 weeks
Change from baseline in the evaluation of the tolerance (excellent, good, average, bad) at 6 weeks | baseline and after 6 weeks
Change from baseline in the evaluation of the tolerance (excellent, good, average, bad) at 12 weeks | baseline and after 12 weeks
Change from baseline in Beck Depression Inventory score at 6 weeks | baseline and after 6 weeks
Change from baseline in Beck Depression Inventory score at 12 weeks | baseline and after 12 weeks
Change from baseline in visual analogic scales for the global quality of the professional, family life, sleep, fatigue at 6 weeks | baseline and after 6 weeks
Change from baseline in visual analogic scales for the global quality of the professional, family life, sleep,fatigue at 12 weeks | baseline and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Moore, MD, PhD, Study Director — Université Victor Segalen Bordeaux 2
Locations (1):
- Cinical Pharmacology Department - Université Victor Segalen Bordeaux 2, Bordeaux, France

REFERENCES:
- [Background] Malach-Pines A. The Burnout Measure Short version (BMS). International Journal of Stress Management. 2005;12:78-88
- [Background] Benezech M, Mullens E, Lalonde R, Desor D, Messaoudi M. Un anxiolytique naturel : l'hydrolysat trypsique de caséine alpha-s1 de lait bovin. Son intérêt en médecine humaine et vétérinaire. Annales Médico-Psychologiques. 2009;167:605-10.
- [Background] Kim JH, Desor D, Kim YT, Yoon WJ, Kim KS, Jun JS, Pyun KH, Shim I. Efficacy of alphas1-casein hydrolysate on stress-related symptoms in women. Eur J Clin Nutr. 2007 Apr;61(4):536-41. doi: 10.1038/sj.ejcn.1602553. Epub 2006 Nov 29. PMID 17136040
- [Background] Milesi MA, Lacan D, Brosse H, Desor D, Notin C. Effect of an oral supplementation with a proprietary melon juice concentrate (Extramel) on stress and fatigue in healthy people: a pilot, double-blind, placebo-controlled clinical trial. Nutr J. 2009 Sep 15;8:40. doi: 10.1186/1475-2891-8-40. PMID 19754931
- [Background] Kong WX, Chen SW, Li YL, Zhang YJ, Wang R, Min L, Mi X. Effects of taurine on rat behaviors in three anxiety models. Pharmacol Biochem Behav. 2006 Feb;83(2):271-6. doi: 10.1016/j.pbb.2006.02.007. Epub 2006 Mar 15. PMID 16540157
- [Background] Facchinetti F, Neri I, Tarabusi M. Eleutherococcus senticosus reduces cardi-ovascular stress response in healthy subjects: a randomized, placebo-controlled trial. Stress and Health. 2002;18:11-7.
- [Background] Hartz AJ, Bentler S, Noyes R, Hoehns J, Logemann C, Sinift S, Butani Y, Wang W, Brake K, Ernst M, Kautzman H. Randomized controlled trial of Siberian ginseng for chronic fatigue. Psychol Med. 2004 Jan;34(1):51-61. doi: 10.1017/s0033291703008791. PMID 14971626